CLINICAL TRIAL: NCT02471963
Title: Randomized, Double-blind, Placebo Controlled, Crossover Clinical Study to Analyse the Effect of Empagliflozin on Macrovascular and Microvascular Circulation and on Endothelium Function
Brief Title: Effect of Empagliflozin on Macrovascular and Microvascular Circulation and on Endothelium Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med. Roland E. Schmieder, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRC2014EMPA
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Empagliflozin; Diabetes mellitus; Macro- and Microcirculation; Vascular Improvement; Endothelium function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin, 25 mg/day, oral administration, 6 weeks
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo, oral administration, 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Empagliflozin may lead to improved vascular and endothelial function in the macro- (pulse wave reflection) and microcirculation (retinal circulation) and improve cardiovascular risk factors, imparticular by effectively controlling hyperglycemia, arterial hypertension and obesity.

DETAILED DESCRIPTION:
Diabetes mellitus, considered as a metabolic disorder, mutates into a predominantly vascular disease, once its duration extends over several years and/or when additional cardiovascular risk factors coexists, in particular arterial hypertension. In accordance, patients with type 2 diabetes die because of microvascular and macrovascular complications, and only rarely because of hypoglycaemic or hyperglycaemic shock syndromes. As a consequence, treatment of type 2 diabetes should focus not only on metabolic control but also on improving the global vascular risk. Analyses that have compared the importance of the various cardiovascular risk factors concluded that reductions of blood pressure and lipid levels are significantly more important than reduction of hyperglycemia. Of course, a multidisciplinary approach is desirable and the STENO-2 study has clearly indicated that in mid-term microvascular complications and in long-term macrovascular complications can be prevented in type 2 diabetes.

Vascular changes occurring in the course of type 2 diabetes, arterial hypertension and elevated global cardiovascular risk can now reliably assessed non-invasively, and already at the very early stage of vascular remodeling processes. For example, the guidelines of the European Society of Hypertension recommend several vascular parameters to be assessed already at the diagnosis of the disease in order to analyze early organ damage of the arteries. The measurement of pulse wave velocity, pulse wave analysis, central (aortic) systolic pressure and pulse pressure are tools to detect early vascular changes in the large arteries related to a faster wave reflection in the arterial tree. Wall to lumen ratio of retinal arteries, retinal capillary flow and flow mediated vasodilation are tools to detect changes in the microvascular circulation. These parameters are only infrequently measured in studies with type 2 diabetes, mainly due to lack of awareness that the vascular changes are the key prognostic factor in type-2 diabetes that ultimately determine the fate of the patient.

Empagliflozin is a novel selective SLGT-2 inhibitor that has been shown to improve glycaemic control after 2, 12, and 24 weeks as well as after 1 and 2 years. Empagliflozin produced dose dependent increases in glucosuria and clinically meaningful changes of glycemic parameters in type 2 diabetes in addition to weight loss. Most striking, empagliflozin was also found to lower systolic blood pressure by 5 mmHg. This reduction in blood pressure might be related to weight loss or/and concomitant loss of total body sodium content. However, the precise mechanism of the blood pressure reduction needs to be elucidated. Loss of sodium would lead to a less reactive contraction of the small arteries in response to increased sympathetic activity, angiotensin II and catecholamines.

Moreover, the endothelium dependent vasodilation after reactive hyperemia is a new non-invasive tool to detect changes on the organ perfusion level. To further assess flow-mediated/Endothelium dependent vasodilation we can assess the EndoPAT Risk Score.

These parameters are only infrequently measured in studies with type 2 diabetes, mainly due to the lack of expertise required to assess these vascular parameters and lack of awareness that vascular changes are the key prognostic factor in type 2 diabetes (and not glycosylated hemoglobin).

In summary, empagliflozin exert beneficial effects on a variety of cardiovascular risk factors, such as hyperglycaemia, hypertension and obesity. These changes should lead (so the hypothesis) to improved vascular and endothelial function in the micro- and macrocirculation.

However, the latter is nothing more than hypothesis and requires clear proof by clinical studies in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus defined by fasting glucose ≥ 126 mg/dl or HbA1c ≥ 6.5% or on blood glucose lowering medication
* Age of 18 - 75 years
* Male and Female patients (females of child bearing potential must be using adequate contraceptive precautions)
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit
* Informed consent (§ 40 Abs. 1 Satz 3 Punkt 3 AMG) has to be given in written form.

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Use of insulin, glitazone, gliptine or SGLT-2 inhibitor within the past 3 months
* Patients with more than one oral blood glucose lowering medication
* Any other oral antidiabetic drug that cannot be discontinued for the study period
* HbA1c ≥ 10%
* Fasting plasma glucose > 240 mg/dl
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 6 months prior to study inclusion
* UACR ≥ 300 mg/g (early morning spot urine)
* eGFR < 60 ml/min/1.73m²
* Uncontrolled arterial hypertension (RR ≥ 180/110 mmHg)
* Congestive heart failure (CHF) NYHA stage III and IV
* Severe disorders of the gastrointestinal tract or other diseases which interfere the pharmacodynamics and pharmakinetics of study drugs
* Significant laboratory abnormalities such as SGOT or SGPT levels more than 3 x above the upper limit of normal range
* Drug or alcohol abusus
* Pregnant or breast-feeding patients
* Use of loop diuretics
* History of repetitive urogenital infection per year
* Body mass index > 40 kg/m²
* Triglyceride levels > 1000 mg/dl
* HDL-cholesterol levels < 25 mg/dl
* Any patient currently receiving chronic (>30 consecutive days) treatment with an oral corticosteroid
* History of epilepsia or history of seizures
* Patients being treated for severe auto immune disease e.g. lupus
* Participation in another clinical study within 30 days prior to visit 1
* Individuals at risk for poor protocol or medication compliance
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Effect of empagliflozin after 6 weeks of treatment on macrocirculation | 6 weeks
  To analyse the effect of empagliflozin after 6 weeks of treatment on macrocirculation as assessed by the pulse wave reflection in the peripheral arterial tree with the composite parameters: central (aortic) systolic pressure, central (aortic) pulse pressure, augmentation pressure, forward wave amplitude, backward wave amplitude and the ratio of forward and backward (pulse wave velocity) compared to placebo.

SECONDARY OUTCOMES:
Effect of empagliflozin after 6 weeks of treatment on microcirculation | 6 weeks
  To analyse the effect of empagliflozin after 6 weeks of treatment on retinal capillary flow (as key measurement of vascular remodeling in the microcirculation) and retinal vascular structural components.
Endothelium Function | 6 weeks
  To analyse the effect of empagliflozin after 6 weeks of treatment on peripheral endothelial function by measuring endothelium-mediated changes in arterial tone using a reactive hyperemia procedure
Biomarkers | 6 weeks
  To analyse the effect of empagliflozin after 6 weeks of treatment on biomarkers for inflammation, metabolic disorders and albuminuria.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof., Principal Investigator — Department of Medicine 4, University of Erlangen-Nuernberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Result] Striepe K, Jumar A, Ott C, Karg MV, Schneider MP, Kannenkeril D, Schmieder RE. Effects of the Selective Sodium-Glucose Cotransporter 2 Inhibitor Empagliflozin on Vascular Function and Central Hemodynamics in Patients With Type 2 Diabetes Mellitus. Circulation. 2017 Sep 19;136(12):1167-1169. doi: 10.1161/CIRCULATIONAHA.117.029529. No abstract available. PMID 28923906
- [Derived] Staef M, Ott C, Kannenkeril D, Striepe K, Schiffer M, Schmieder RE, Bosch A. Determinants of arterial stiffness in patients with type 2 diabetes mellitus: a cross sectional analysis. Sci Rep. 2023 Jun 2;13(1):8944. doi: 10.1038/s41598-023-35589-4. PMID 37268640
- [Derived] Gessner A, Gemeinhardt A, Bosch A, Kannenkeril D, Staerk C, Mayr A, Fromm MF, Schmieder RE, Maas R. Effects of treatment with SGLT-2 inhibitors on arginine-related cardiovascular and renal biomarkers. Cardiovasc Diabetol. 2022 Jan 6;21(1):4. doi: 10.1186/s12933-021-01436-x. PMID 34991562
- [Derived] Bosch A, Ott C, Jung S, Striepe K, Karg MV, Kannenkeril D, Dienemann T, Schmieder RE. How does empagliflozin improve arterial stiffness in patients with type 2 diabetes mellitus? Sub analysis of a clinical trial. Cardiovasc Diabetol. 2019 Mar 29;18(1):44. doi: 10.1186/s12933-019-0839-8. PMID 30922297
- [Derived] Kannenkeril D, Bosch A, Harazny J, Karg M, Jung S, Ott C, Schmieder RE. Early vascular parameters in the micro- and macrocirculation in type 2 diabetes. Cardiovasc Diabetol. 2018 Sep 19;17(1):128. doi: 10.1186/s12933-018-0770-4. PMID 30231923